CLINICAL TRIAL: NCT05679453
Title: Comparison of Lornoxicam and Etodolac on Edema, Trismus and Pain After Third Molar Surgery
Brief Title: Lornoxicam Versus Etodolac After Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Zulfikar Karabiyik, Research Assistant, Kutahya Health Sciences University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 10
Record Dates: First submitted 2022-10-31; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Pain, Acute; Edema; Trismus
MeSH Terms: conditions — Acute Pain; Edema; Trismus | interventions — lornoxicam; Tablets; Etodolac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etodolac (Active Comparator): Etodolac, 400 mg tid per a day for four days
  Interventions: Drug: Lornoxicam 8 Mg Oral Tablet
- Lornoxicam (Active Comparator): Lornoxicam, 8 mg twice per day for four days
  Interventions: Drug: Lornoxicam 8 Mg Oral Tablet

INTERVENTIONS:
Drug: Lornoxicam 8 Mg Oral Tablet — Lornoxicam is a oxicam grup non-steroid antiinflamatuar drug
  Other Names: Etodolac

SUMMARY:
Our study aimed to compare the effect of lornoxicam and etodolac on postoperative pain, edema and trismus following lower third molar extraction

DETAILED DESCRIPTION:
20 patients included in study (4 male, 16 female). Lornoxicam and etodolac was given following lower third molar extraction. Pain was evaluated 2., 6., 12., 24., and 48. hours using VAS. Edema was evaluated by measuring tragus-labial commissure, angulus- lateral canthus of eye and angulus mandible-labial commissure. Trismus was evaluated measuring mouth opening by caliper. Edema and Trismus was evaluated by 48. and 168. hours

ELIGIBILITY:
Inclusion Criteria:

* Bilateral mesioangular impacted lower third molar
* Asymptomatic Third Molar (No history of infection)
* Systemically Healthy Person
* Person Between aged 18-30

Exclusion Criteria:

* People who are pregnant and lactation process
* People who had any systemic disease
* People who are gastrointestinal problems
* People who are sensitive to drugs used in study
* Lower Third Molar associated with cysts and infections

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Pain after wisdom tooth extraction | 2 th hours
  Pain after lower third molar removal, Pain was evaluated with VAS(visual anolog scale)
Edema after wisdom tooth extraction | 48 th hours
  Edema lower third molar removal, Edema was evaluated by using reference line on the face
Trismus after wisdom tooth extraction | 48 th hours,
  Trismus lower third molar removal, trismus was evaluated by using caliper

SECONDARY OUTCOMES:
Pain after wisdom tooth extraction | 6 th hours
  Pain after lower third molar removal, Pain was evaluated with VAS(visual anolog scale)
Pain after wisdom tooth extraction | 12 th hours
  Pain after lower third molar removal, Pain was evaluated with VAS(visual anolog scale)
Pain after wisdom tooth extraction | 24 th hours
  Pain after lower third molar removal, Pain was evaluated with VAS(visual anolog scale)
Pain after wisdom tooth extraction | 48 th hours
  Pain after lower third molar removal, Pain was evaluated with VAS(visual anolog scale)
Edema after wisdom tooth extraction | 168 th hours
  Edema lower third molar removal, Edema was evaluated by using reference line on the face
Trismus after wisdom tooth extraction | 168 th hours
  Trismus lower third molar removal, trismus was evaluated by using caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Zülfikar Karabıyık, Kütahya, Turkey (Türkiye)